CLINICAL TRIAL: NCT02813577
Title: A Prospective, Multicenter, Single Arm, Post-Approval Study of the Lutonix Drug Coated Balloon for Treatment of Femoropopliteal Arteries in United States Females
Brief Title: Lutonix Drug Coated Balloon for Treatment of Femoropopliteal Arteries in United States Females (CONFIRM)
Acronym: CONFIRM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: FDA allowed other data to be leveraged to meet the study requirements
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL0025-01
Record Dates: First submitted 2016-06-16; First posted 2016-06-27 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Femoral Artery Stenosis; Popliteal Artery Stenosis; Femoral Artery Occlusion; Popliteal Artery Occlusion
Keywords: Legs; Drug Coated Angioplasty Balloon; Experimental; Standard Angioplasty Balloon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Lutonix® 035 Drug Coated Balloon PTA Catheter (Other): This is a single-arm study. Female subjects will receive the Lutonix® 035 Drug Coated Balloon PTA Catheter.
  Interventions: Device: Lutonix® 035 Drug Coated Balloon PTA Catheter

INTERVENTIONS:
Device: Lutonix® 035 Drug Coated Balloon PTA Catheter — Female subjects will receive the Lutonix® 035 Drug Coated Balloon PTA Catheter.

SUMMARY:
The post approval study will enroll US female patients presenting with claudication or ischemic rest pain and an angiographically significant lesion in the superficial femoral or popliteal artery. Subjects are treated per Instructions For Use (IFU) with the Lutonix® Catheter. Subjects will have a Duplex Ultrasound (DUS) and clinical follow-up through two (2) years.

DETAILED DESCRIPTION:
The Lutonix® 035 Drug Coated Balloon PTA Catheter (Lutonix® Catheter) has been approved by the Food and Drug Administration (P130024) for percutaneous transluminal angioplasty, after appropriate vessel preparation of de novo, restenotic, or in-stent restenotic lesions up to 300 mm in length in native superficial femoral or popliteal arteries with reference vessel diameters of 4-7 mm. The purpose of this post-approval study is to assess the safety and effectiveness of the Lutonix® Catheter in the US female population. This study will enroll approximately 165 female patients at a minimum of 10 US centers and a maximum of 25.

ELIGIBILITY:
Clinical Criteria

1. Non-pregnant female ≥18 years of age;
2. Rutherford Clinical Category 2-4;
3. Patient is willing to provide informed consent, is geographically stable, comply with the required follow up visits and testing schedule;

   Angiographic Criteria
4. De novo or restenotic lesion(s) in native superficial femoral or popliteal arteries;
5. Lesion ≥70% stenosis by visual estimate;
6. Target reference vessel diameter of 4-7 mm;
7. A patent inflow artery free from significant lesion (≥50% stenosis) as confirmed by angiography; (Treatment of target lesion acceptable after successful treatment of inflow artery lesions. Successful inflow artery treatment is defined as attainment of residual diameter stenosis ≤30% without death or major vascular complication.)
8. At least one patent native outflow artery to the ankle, free from significant (≥50%) stenosis as confirmed by angiography after successful vessel preparation;
9. Successful antegrade wire crossing and vessel preparation (may include pre-dilatation) of the target lesion. Successful vessel preparation is defined by residual stenosis ≤30% without any major vascular complications;
10. No other prior vascular interventions within 2 weeks before and/or planned 30 days after the protocol treatment except for remote common femoral patch angioplasty separated by at least 2 cm from the lesion(s).

Exclusion Criteria

1. Life expectancy of <2 years;
2. Subject is currently participating in an investigational drug or device study, or previously enrolled in this study. Enrollment in another investigational drug or device study during the follow up period is not allowed;
3. History of stroke within 3 months;
4. History of myocardial infarction (MI), thrombolysis or angina within 2 weeks of index procedure;
5. Renal failure or chronic kidney disease with serum creatinine ≥2.5 mg/L within 30 days of index procedure or treated with dialysis;
6. Sudden symptom onset, acute vessel occlusion, or acute or sub-acute thrombus in target vessel.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2019-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Metzger, MD, Principal Investigator — Wellmont CVA Heart Institute
Locations (4):
- United States (4):
  - St. Vincent Medical Group, Indianapolis, Indiana
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - Vascular Access Solutions, Orangeburg, South Carolina
  - Wellmont CVA Heart Institute, Kingsport, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Lutonix® 035 Drug Coated Balloon PTA Catheter Instructions For Use — http://www.bardpv.com/?portfolio=lutonix-035

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lutonix® 035 Drug Coated Balloon PTA Catheter
Started | 4
Completed | 0 (Study was terminated and only some results at 1 month follow up are available.)
Not Completed | 4
Not completed — Study terminated | 4

BASELINE CHARACTERISTICS:
Arm/Group | Lutonix® 035 Drug Coated Balloon PTA Catheter
Number analyzed (Participants) | 4
Age, Customized [Count of Participants; unit: Participants]
  ≥18 years of age | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Freedom From the Following: All-cause Peri-operative Death at 30 Days, Index Limb Amputation Within 1 Year, Index Limb Re-intervention Within 1 Year, and Index-limb-Related Death Within 1 Year Post Index Procedure
Description: Index limb amputation includes above or below the ankle amputations.
Time Frame: 12 months post index procedure
Population: Study was terminated.
Arm/Group | Lutonix® 035 Drug Coated Balloon PTA Catheter
Number analyzed (Participants) | 0

2. Primary Outcome: Effectiveness: Number of Participants With Primary Patency of the Target Lesion at 12 Month Post Index Procedure.
Description: Primary patency is defined as freedom from target lesion restenosis (TLR) and from binary restenosis. Binary restenosis is adjudicated by the independent Core Laboratory based on Peak Systolic Velocity Ratio (PSVR) ≥ 2.5 and / or abnormal waveforms, or based on angiographic ≥ 50% diameter stenosis.
Time Frame: 12 months post index procedure
Population: Study was terminated.
Arm/Group | Lutonix® 035 Drug Coated Balloon PTA Catheter
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Freedom From All-cause Perioperative (≤ 30 Day) Death and Freedom From the Following: Index Limb Amputation, Index Limb Re-intervention, and Index-Limb-Related Death.
Time Frame: 30 days post index procedure
Population: Study was terminated.
Arm/Group | Lutonix® 035 Drug Coated Balloon PTA Catheter
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Major Vascular Complications at 30 Days Post Index Procedure
Time Frame: 30 days
Measure: Number; unit: Complications
Arm/Group | Lutonix® 035 Drug Coated Balloon PTA Catheter
Number analyzed (Participants) | 4
Complications | 0

5. Secondary Outcome: Number of Deaths (All Causes) at 30 Days Post Index Procedure
Time Frame: 30 days post index procedure
Measure: Number; unit: Participants
Arm/Group | Lutonix® 035 Drug Coated Balloon PTA Catheter
Number analyzed (Participants) | 4
Participants | 0

6. Secondary Outcome: Number of Participants With Clinically Driven Target Lesion Revascularization (TLR) at 1, 6, 12, and 24 Month Post Index Procedure
Time Frame: 1, 6, 12 and 24 months post index procedure
Population: Study terminated.
Arm/Group | Lutonix® 035 Drug Coated Balloon PTA Catheter
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR) at 1, 6, 12, and 24 Months Post Index Porcedure
Time Frame: 1, 6, 12 and 24 months post index procedure
Population: Study was terminated.
Arm/Group | Lutonix® 035 Drug Coated Balloon PTA Catheter
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Participants With Reintervention for Treatment of Thrombosis of the Target Vessel or Embolization to Its Distal Vasculature at 1, 6, 12, and 24 Months Post Index Procedure
Time Frame: 1, 6, 12 and 24 months post index procedure
Population: Study was terminated.
Arm/Group | Lutonix® 035 Drug Coated Balloon PTA Catheter
Number analyzed (Participants) | 0

9. Secondary Outcome: Number of Participants With Unanticipated and Anticipated Device Related Serious Adverse Events at 1, 6, 12, and 24 Months Post Index Procedure
Time Frame: 1, 6, 12 and 24 months post index procedure
Population: Study was terminated.
Arm/Group | Lutonix® 035 Drug Coated Balloon PTA Catheter
Number analyzed (Participants) | 0

10. Secondary Outcome: Number of Participants With Amputation (Above the Ankle)-Free Survival (AFS) at 1, 6, 12, and 24 Months Post Index Procedure.
Time Frame: 1, 6, 12 and 24 months
Population: Study was terminated.
Arm/Group | Lutonix® 035 Drug Coated Balloon PTA Catheter
Number analyzed (Participants) | 0

11. Secondary Outcome: Change in Rutherford Classification Scores at 1, 6, 12, and 24 Months Post Index Procedure Compared to Baseline
Time Frame: 1, 6, 12 and 24 months post index procedure
Population: Study was terminated.
Arm/Group | Lutonix® 035 Drug Coated Balloon PTA Catheter
Number analyzed (Participants) | 0

12. Secondary Outcome: Number of Participants With Sustained Clinical Benefit at 1, 6, 12, and 24 Months Post Index Procedure
Time Frame: 1, 6, 12 and 24 months post index procedure
Population: Study was terminated.
Arm/Group | Lutonix® 035 Drug Coated Balloon PTA Catheter
Number analyzed (Participants) | 0

13. Secondary Outcome: Change of Resting Ankle Brachial Index (ABI) Scores at 1, 6, 12, and 24 Months Post Index Procedure Compared to Baseline
Time Frame: 1, 6, 12 and 24 months post index procedure
Population: Study was terminated.
Arm/Group | Lutonix® 035 Drug Coated Balloon PTA Catheter
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: At 1 month post-index procedure.
Description: Only the following type of endpoint related adverse events were reported:
  * Events leading to death
  * Target limb reintervention
  * Target limb amputation
  * Any event deemed to be device- or procedure-related
  * Major vascular complication within 30 days of the index procedure
  * Any event involving the target limb that requires treatment
Arm/Group | Lutonix® 035 Drug Coated Balloon PTA Catheter
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to PI publication of site results, sponsor requires publication of multi-centers results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT02813577/Prot_SAP_000.pdf